CLINICAL TRIAL: NCT01321606
Title: IMpact of PRObiotics for Reducing Infections in VEterans: The IMPROVE Study
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Collaborators: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: CLIN-010-10S; OMB 4040-0001 (Other: University of Wisconsin, Madison)
Record Dates: First submitted 2011-03-21; First posted 2011-03-23 (Estimated); Results first posted 2018-08-03 (Actual); Last update posted 2018-08-03 (Actual); Status verified 2017-11

CONDITIONS: Anti-biotic Resistance
Keywords: infection; probiotics
MeSH Terms: conditions — Infections | interventions — Sugars

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm 1: Probiotic (Experimental): subjects will be given a capsule formulation of a 1x10^10 colony-forming units of probiotic L. rhamnosus HN001 to be taken once a day, for 4 weeks
  Interventions: Dietary Supplement: Lactobacillus rhamnosus HN001
- Arm 2: Placebo (Placebo Comparator): Placebo identical to the active product will be given
  Interventions: Dietary Supplement: sugar pill (placebo)

INTERVENTIONS:
Dietary Supplement: Lactobacillus rhamnosus HN001 — Subjects will be given a pill formulation of a probiotic L. rhamnosus HN001 to be taken once a day, at a dose of 1 x 10^10 organisms
  Arms: Arm 1: Probiotic
Dietary Supplement: sugar pill (placebo) — Placebo identical to the active product will be given
  Arms: Arm 2: Placebo

SUMMARY:
The investigators have two hypotheses: (1) The probiotic L. rhamnosus HN001, when compared to placebo, will reduce S. aureus nasal colonization when taken for four weeks. (2) The probiotic L. rhamnosus HN001, when compared to placebo, will reduce S. aureus gastrointestinal colonization when taken for four weeks.

DETAILED DESCRIPTION:
Reducing infections caused by S. aureus is essential. The knowledge that colonization at a few key body sites such as the nose and the gastrointestinal tract is a prerequisite for infection2 ,3 offers an opportunity for therapeutic intervention. Thirty percent of the population has nasal colonization with S. aureus. In the last few years, decolonization agents such as mupirocin topical ointment and oral antibiotics such as doxycycline and rifampin have been studied for their utility in reducing colonization. However, these options have limitations in that recolonization is common, the impact of these interventions on multiple sites of colonization has not been assessed and resistance develops frequently to any of these, especially the oral antibiotics. Resistance in S. aureus has been designated a public health crisis. Methicillin-resistant S. aureus (MRSA) now accounts for 60% of all S. aureus infections. As an example of the growing crisis in S. aureus resistance, it should be noted that the number of MRSA infections rose from 2000 in 1993 to 368,000 in 2005. MRSA infections pose an even greater health and economic burden on the population than those caused by methicillin-sensitive S. aureus.4-8 S. aureus and MRSA infection trends in the VA health system mirror national trends5 and are associated with considerable morbidity and mortality in Veterans. A treatment that reduces S. aureus and MRSA colonization, without a risk of promoting antibiotic resistance could represent a breakthrough in decolonization therapy. Probiotics may be one such treatment option.

Probiotics are live microorganisms that are available over the counter, widely used as dietary supplements or nutritional foods and represent a low-cost, well tolerated, safe, non-antibiotic based strategy that may have efficacy for decolonization without the attendant risks of promoting antimicrobial resistance.9 Certain probiotics, including Lactobacillus rhamnosus HN001, have demonstrated ability to stimulate systemic immune functions, possibly enhancing the body's ability to eradicate S. aureus in the gastrointestinal tract and at sites remote from the gastrointestinal tract such as the nose.10 ,11 The long-term goal of this research is to identify and test novel interventions for reducing infections caused by resistant bacteria. The investigators propose a Phase II randomized, double-blind, placebo-controlled clinical trial in Veterans to evaluate the efficacy of an oral probiotic, Lactobacillus rhamnosus HN001, for reducing S. aureus colonization. This study will produce data, methods, and tools that have widespread relevance and portability, with the potential to reduce healthcare-associated infections.

ELIGIBILITY:
Inclusion Criteria:

* Colonized at nasal or gastrointestinal source by S. aureus including MRSA
* Age 18 years or older
* Able to take oral medications
* Able to provide informed consent

Exclusion Criteria:

Uncontrolled psychiatric illness

* On a decolonization protocol for MRSA (e.g mupirocin, tea tree oil)
* Current involvement in another investigational trial
* Pregnancy
* Persistent diarrhea (> 3 loose stools per day for at least 2 days)
* Active infection with S.aureus or MRSA

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 113 (Actual)
Dates: Start 2011-10; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nasia Safdar, MD PhD, Principal Investigator — William S. Middleton Memorial Veterans Hospital, Madison, WI
Locations (1):
- William S. Middleton Memorial Veterans Hospital, Madison, WI, Madison, Wisconsin, United States

REFERENCES:
- [Derived] Eggers S, Barker AK, Valentine S, Hess T, Duster M, Safdar N. Effect of Lactobacillus rhamnosus HN001 on carriage of Staphylococcus aureus: results of the impact of probiotics for reducing infections in veterans (IMPROVE) study. BMC Infect Dis. 2018 Mar 14;18(1):129. doi: 10.1186/s12879-018-3028-6. PMID 29540160
- [Derived] Eggers S, Barker A, Valentine S, Hess T, Duster M, Safdar N. Impact of Probiotics for Reducing Infections in Veterans (IMPROVE): Study protocol for a double-blind, randomized controlled trial to reduce carriage of Staphylococcus aureus. Contemp Clin Trials. 2017 Jan;52:39-45. doi: 10.1016/j.cct.2016.11.004. Epub 2016 Nov 9. PMID 27836508

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm 1a: Extra-GI Probiotic: Subjects with Extra-GI colonization at initial screening who were randomized to probiotic treatment.
  Extra-GI colonization was defined as a positive PCR result for S. aureus from any swab of the nares, axillae or wound, with no positive result from swabs of the oropharynx, or peri-rectum.
  Subjects were given a capsule formulation of a 1x10^10 colony-forming units of probiotic L. rhamnosus HN001 to be taken once a day, for 4 weeks.
- Arm 2a: Extra-GI Placebo: Subjects with Extra-GI colonization at initial screening who were randomized to placebo treatment.
  Extra-GI colonization was defined as a positive PCR result for S. aureus from any swab of the nares, axillae or wound, with no positive result from swabs of the oropharynx, or peri-rectum.
  Placebo pill: composed of identical inactive components to the active product, given to be taken once daily for 4 weeks.
- Arm 1b: GI Probiotic: Subjects with GI colonization at initial screening who were randomized to probiotic treatment.
  GI colonization was defined as a positive PCR result for S. aureus from any swab of the oropharynx, or peri-rectum.
  Subjects were given a capsule formulation of a 1x10^10 colony-forming units of probiotic L. rhamnosus HN001 to be taken once a day, for 4 weeks
- Arm 2b: GI Placebo: Subjects with GI colonization at initial screening who were randomized to placebo treatment.
  GI colonization was defined as a positive PCR result for S. aureus from any swab of the oropharynx, or peri-rectum.
  Placebo pill: composed of identical inactive components to the active product, given to be taken once daily for 4 weeks.
Period: Overall Study
Arm/Group | Arm 1a: Extra-GI Probiotic | Arm 2a: Extra-GI Placebo | Arm 1b: GI Probiotic | Arm 2b: GI Placebo
Started | 18 | 32 | 34 | 29
Completed | 18 | 32 | 34 | 28
Not Completed | 0 | 0 | 0 | 1
Not completed — Lost to Follow-up | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Arm 1: Probiotic: Subjects were given a capsule formulation of a 1x10^10 colony-forming units of probiotic L. rhamnosus HN001 to be taken once a day, for 4 weeks
  Lactobacillus rhamnosus HN001: Subjects will be given a pill formulation of a probiotic L. rhamnosus HN001 to be taken once a day, at a dose of 1 x 10^10 organisms
- Arm 2: Placebo: Placebo composed of identical inactive components to the active product, to be taken once daily for 4 weeks.
  Placebo pill: composed of identical inactive components to the active product, given to be taken once daily for 4 weeks.
- Total: Total of all reporting groups
Arm/Group | Arm 1: Probiotic | Arm 2: Placebo | Total
Number analyzed (Participants) | 52 | 61 | 113
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.4 (14.7) | 62.9 (12.6) | 63.6 (13.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 5 | 8
  Male | 49 | 56 | 105

OUTCOME MEASURES:

1. Primary Outcome: Oral L. Rhamnosus HN001 Therapy Compared to Placebo on Gastrointestinal and Extra-gastrointestinal Colonization of S. Aureus.
Description: Participants in the final outcome may be colonized at both GI and Extra-GI sites, thus the total numbers from the outcome cells can be greater than the overall number of participants analyzed.
Time Frame: 4 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1a: Extra-GI Probiotic | Arm 2a: Extra-GI Placebo | Arm 1b: GI Probiotic | Arm 2b: GI Placebo
Number analyzed (Participants) | 18 | 32 | 34 | 29
Participants
  Endpoint GI colonization | 9 | 17 | 25 | 24
  Endpoint Extra-GI colonization | 16 | 22 | 20 | 19

2. Secondary Outcome: Oral L. Rhamnosus HN001 Therapy Compared With Placebo on Phagocytic Functioning of Polymorphonuclear (PMN) and Monocyte Cells
Description: This outcome is the mean difference in the % of granulocytes that phagocytized E. coli, from blood samples taken at the beginning and end of the trial. Percent of granulocytes phagocytizing E. coli at baseline is subtracted by percent of granulocytes phagocytizing E. coli at the end of the trial. The mean and standard error are calculated and reported for each study arm. This result
Time Frame: 4 weeks
Population: Some participants were excluded from this analysis due to lack of sample collection, or unusable results because tests did not meet acceptability criteria.
Measure: Mean (Standard Error); unit: Difference in % POS of Granulocytes
Arm/Group | Arm 1a: Extra-GI Probiotic | Arm 2a: Extra-GI Placebo | Arm 1b: GI Probiotic | Arm 2b: GI Placebo
Number analyzed (Participants) | 15 | 25 | 27 | 21
Difference in % POS of Granulocytes | -0.29 (2.43) | -1.38 (2.65) | 1.23 (2.42) | 2.61 (2.83)

3. Secondary Outcome: Oral L. Rhamnosus HN001 Therapy Compared With Placebo on Phagocytic Functioning of Polymorphonuclear (PMN) and Monocyte Cells
Description: This outcome is the mean difference in the % of monocytes that phagocytized E. coli, from blood samples taken at the beginning and end of the trial. Percent of monocytes phagocytizing E. coli at baseline is subtracted by percent of monocytes phagocytizing E. coli at the end of the trial. The mean and standard error are calculated and reported for each study arm.
Time Frame: 4 weeks
Population: as for outcome 2
Measure: Mean (Standard Error); unit: Difference in % POS of Monocytes
Arm/Group | Arm 1a: Extra-GI Probiotic | Arm 2a: Extra-GI Placebo | Arm 1b: GI Probiotic | Arm 2b: GI Placebo
Number analyzed (Participants) | 15 | 25 | 27 | 21
Difference in % POS of Monocytes | -0.54 (0.29) | 0.59 (0.32) | 0.07 (0.33) | 0.15 (0.36)

ADVERSE EVENTS:
Time Frame: 4 weeks
Groups:
- Arm 1: Extra-GI Probiotic: Subjects with Extra-GI colonization at initial screening who were randomized to probiotic treatment. Subjects were given a capsule formulation of a 1x10^10 colony-forming units of probiotic L. rhamnosus HN001 to be taken once a day, for 4 weeks
  Lactobacillus rhamnosus HN001: Subjects will be given a pill formulation of a probiotic L. rhamnosus HN001 to be taken once a day, at a dose of 1 x 10^10 organisms
- Arm 2: Extra-GI Placebo: Subjects with Extra-GI colonization at initial screening who were randomized to placebo treatment. Placebo composed of identical inactive components to the active product, to be taken once daily for 4 weeks.
  Placebo pill: composed of identical inactive components to the active product, given to be taken once daily for 4 weeks.
- Arm 3: GI Probiotic: Subjects with GI colonization at initial screening who were randomized to probiotic treatment. Subjects were given a capsule formulation of a 1x10^10 colony-forming units of probiotic L. rhamnosus HN001 to be taken once a day, for 4 weeks
  Lactobacillus rhamnosus HN001: Subjects will be given a pill formulation of a probiotic L. rhamnosus HN001 to be taken once a day, at a dose of 1 x 10^10 organisms
- Arm 4: GI Placebo: Subjects with GI colonization at initial screening who were randomized to placebo treatment. Placebo composed of identical inactive components to the active product, to be taken once daily for 4 weeks.
  Placebo pill: composed of identical inactive components to the active product, given to be taken once daily for 4 weeks.
Arm/Group | Arm 1: Extra-GI Probiotic | Arm 2: Extra-GI Placebo | Arm 3: GI Probiotic | Arm 4: GI Placebo
Serious Adverse Events (participants affected / at risk) | 0/18 | 2/32 | 0/34 | 0/29
Other Adverse Events (participants affected / at risk) | 9/18 | 17/32 | 17/34 | 14/29
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1: Extra-GI Probiotic (N=18) | Arm 2: Extra-GI Placebo (N=32) | Arm 3: GI Probiotic (N=34) | Arm 4: GI Placebo (N=29)
Cardiovascular event (Cardiac disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Arm 1: Extra-GI Probiotic (N=18) | Arm 2: Extra-GI Placebo (N=32) | Arm 3: GI Probiotic (N=34) | Arm 4: GI Placebo (N=29)
Fever (General disorders) | 0 | 2 | 1 | 1
Nausea/Vomiting (Gastrointestinal disorders) | 3 | 5 | 4 | 2
Constipation (Gastrointestinal disorders) | 4 | 2 | 0 | 1
Cough/Cold/Congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 5 | 3 | 6
Muscle Pain/Cramp/Spasm (Musculoskeletal and connective tissue disorders) | 3 | 5 | 11 | 4
Upset Stomach/Heartburn (Gastrointestinal disorders) | 1 | 1 | 1 | 1
Gas/Bloating (Gastrointestinal disorders) | 2 | 1 | 1 | 1
Unusual Stool (Gastrointestinal disorders) | 2 | 8 | 7 | 5
Bad Taste (General disorders) | 0 | 2 | 0 | 1
Itchiness (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No